CLINICAL TRIAL: NCT05667454
Title: Investigator Led, Double-masked, Multicenter, Randomized Clinical Trial for the Comparison of Atropine 0.5% Versus Atropine 0.05% Eye Drops for the Prevention of Myopia Progression in Dutch Children
Brief Title: MAD Trial: Myopia Atropine Dose
Acronym: MAD
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Principal Investigator, Caroline C.W. Klaver, MD, Prof. dr. C.C.W. Klaver, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NL78526.078.21; MEC-2021-0814 (Other: METC Erasmus MC); 2021-004015-11 (EudraCT Number)
Record Dates: First submitted 2022-11-21; First posted 2022-12-28 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Progressive Myopia
Keywords: Myopia; Atropine; Axial length; Child
MeSH Terms: conditions — Myopia, Degenerative; Myopia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Low dose atropine (Active Comparator): Atropine 0.05% sulphate ophthalmic solution should be administered, one drop in each eye, once daily, at bedtime, for 3 years.
  Interventions: Drug: Atropine Ophthalmic 0.05%
- High dose atropine (Active Comparator): Atropine 0.5% sulphate ophthalmic solution should be administered, one drop in each eye, once daily, at bedtime, for 3 years.
  Interventions: Drug: Atropine Ophthalmic 0.5%

INTERVENTIONS:
Drug: Atropine Ophthalmic 0.05% — Atropine 0.05% sulphate ophthalmic solution
  Arms: Low dose atropine
Drug: Atropine Ophthalmic 0.5% — Atropine 0.5% sulphate ophthalmic solution
  Arms: High dose atropine

SUMMARY:
The goal of this interventional study is to compare the efficacy of Atropine 0.05% to Atropine 0.5% treatment against progression of axial length in European children with progressive myopia, and to evaluate the safety, adherence, and reasons for nonresponse. Subjects will use Atropine eye drops for a period of 3 years, followed by a 2 year observational period.

DETAILED DESCRIPTION:
With the current worldwide myopia boom the frequency of high myopia will also increase, and potentially blinding complications such as myopic macular degeneration, retinal detachment, and glaucoma will occur more often. In the Netherlands high myopia will become the most important cause of low vision and blindness by 2050. As treatment options are limited once the eye is fully grown, prevention of a long axial length at childhood is the only way to counteract this prospect. Pharmacological interventions have shown a high efficacy in stopping eye growth, in particular eye drops with high dose Atropine (0.5%, 1%). Nevertheless, the high frequency of side effects (photophobia, reading problems) of these Atropine concentrations has favoured the use of low dose Atropine. Atropine 0.01% is the most commonly used and lowest dosage; it has shown stability of refractive error, but not of axial length. Recent studies have shown that Atropine 0.05% has low risk of side effects, but a higher efficacy than 0.01%. Many ongoing trials are now comparing various low dose Atropine to placebo, but none are comparing the highest low dose to the lowest high dose Atropine.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6 to ≤ 11 years with bilateral myopia
* Onset of myopia ≥ 4 years of age
* History of progression
* SER of at least -1.00D and no greater than -6.00D in each eye measured using cycloplegic auto refraction
* Intraocular pressure < 21 mm Hg in each eye
* Distance vision correctable to at least 0.1 Log MAR (logarithm of the minimum angle of resolution) in each eye

Exclusion Criteria:

* Allergy to atropine or other excipients of the eye drops
* History of amblyopia or strabismus
* History of retinal dystrophy or systemic disorder
* Abnormal ocular biometry aside from axial length
* History of glaucoma
* Chronic use of topical or systemic antimuscarinic/anticholinergic medications in the 21 days prior to screening, and/or anticipated need for chronic use over the duration of the study (i.e., more than 7 consecutive days in 1 month or more than a total of 30 days in 1 year).
* Chronic use (more than 3 days a week) of topical ophthalmological medication (prescribed or over the counter) other than the assigned study medication. The use of artificial tears is allowed but not in the 1 hour before or after the administration of the study medication.
* The anticipated need to use chronic ophthalmic or systemic oral corticosteroids during the study. (i.e., < 2 weeks)
* Prior myopia treatments.
* Employees of the study center and their family members.

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 550 (Estimated)
Dates: Start 2022-12-19 (Actual); Primary Completion 2029-03-01 (Estimated); Study Completion 2029-04-01 (Estimated)

PRIMARY OUTCOMES:
Progression of axial length in mm from baseline to t = 36 months. | 3 years

SECONDARY OUTCOMES:
Progression of axial length in mm from baseline to t = 60 months. | 5 years
Progression of spherical equivalent of refraction in dioptres from baseline to t = 36 months. compared to atropine 0.5% treatment. | 3 years
Progression of spherical equivalent of refraction in dioptres from baseline to t = 60 | 5 years
Proportion of subjects who show ≤ 0.20 mm (good response); 0.2 - 0.3 mm (acceptable response), and > 3 mm (nonresponse) | 3 years
Proportion of subjects who progressed to high myopia (AL 26+ mm) | 3 years
Change in visual function (BCVA, contrast sensitivity, and glare) | 3 years
Frequency and type of treatment-related (serious) adverse events as assessed by CTCAE v5.0 (=safety) | 3 years
Proportion of non-adherence | 3 years
Difference in health related quality of life | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: C.C.W. Klaver, Prof. Dr., Principal Investigator — EMC
Locations (20):
- Netherlands (20):
  - Flevoziekenhuis, Almere Stad
  - OLVG, locatie Oost, Amsterdam
  - Ophthalmologistenpraktijk Delfland, Delft
  - Reinier de Graaf Gasthuis, Delft
  - Deventer Ziekenhuis, Deventer
  - Albert Schweitzer ziekenhuis, Dordrecht
  - Bergman Clinics - Ede, Ede
  - Admiraal de Ruyter Ziekenhuis, Goes
  - Frisius MC, Heerenveen
  - Oogcentrum Noordholland, Heerhugowaard
  - Leiden University Medical Center, Leiden
  - Bergman Clinics - Lelystad, Lelystad
  - Maastricht UMC+, Maastricht
  - St. Antonius, Nieuwegein
  - Radboudumc, Nijmegen
  - Erasmus Medical Center, Rotterdam
  - Haga Ziekenhuis, The Hague
  - Oogkliniek Den Haag, The Hague
  - Ziekenhuis Rivierenland Tiel, Tiel
  - Elisabeth-TweeSteden Ziekenhuis, Tilburg

IPD SHARING:
Plan to Share IPD: Undecided